CLINICAL TRIAL: NCT06128993
Title: Trans-coronary Cooling and Dilution for Cardioprotection During Revascularisation for ST-elevation Myocardial Infarction
Acronym: STEMI-Cool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 315559
Record Dates: First submitted 2023-10-17; First posted 2023-11-13 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-11

CONDITIONS: Myocardial Infarction; Reperfusion Injury, Myocardial
MeSH Terms: conditions — Myocardial Infarction; Myocardial Reperfusion Injury | interventions — Indicator Dilution Techniques; Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomised placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcoronary cooling and dilution (Experimental): Intervention with transcoronary cooling and dilution
  Interventions: Other: Transcoronary cooling and dilution
- Standard of care (Active Comparator): Routine clinical care
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Transcoronary cooling and dilution — Transcoronary cooling and dilution
  Arms: Transcoronary cooling and dilution
Other: Standard of care — Routine clinical care
  Arms: Standard of care

SUMMARY:
A heart attack (myocardial infarction) occurs when an artery supplying blood to the heart is suddenly blocked resulting in damage to the heart muscle.

Patients presenting to hospital with a heart attack undergo an immediate angiogram (x-ray of the arteries in the heart) and are usually treated immediately with a balloon and stent to open their blocked artery. This procedure is called "primary percutaneous coronary intervention" (or primary PCI for short).

An angiogram is a routine procedure that involves insertion of fine plastic tube (catheter) into either the groin or wrist under local anaesthetic. The tube is passed into the artery in the heart and X-ray pictures are taken to find out if the arteries are blocked. Blocked arteries can usually be opened by passing a small balloon into the artery, via the fine plastic tube followed by placement of a stent (a fine metal coil) into the artery to prevent it from blocking again.

Although this treatment is very successful, it can result in damage to the heart muscle when the artery is opened. Cooling the entire body has been shown to reduce heart muscle damage during heart attacks in some patients but not in others; however, it is uncomfortable due to the shivering, expensive and can result in delays in opening the blocked artery.

The investigators are conducting a series of research studies to find out if cooling the heart muscle directly through the catheter being used for the normal primary angioplasty treatment using room temperature may be effective in preserving heart muscle, without the shortcomings of entire body cooling.

The investigators have already published an initial series of ten cases in which this treatment appeared to be feasible without causing significant clinical problems.

The present study is a pilot study designed to assess the rate of patient recruitment and feasibility of this new treatment while exploring some detailed outcomes measuring the restoration of blood flow within the coronary artery at the end of the procedure.

Ultimately if the present pilot study is successful, the investigators plan to go on to undertake a much larger randomised outcome study to determine definitively whether this treatment can help reduce heart attack size.

DETAILED DESCRIPTION:
The study population will comprise 60 patients with ST-Elevation Myocardial Infarction (STEMI) presenting to Harefield Hospital undergoing primary percutaneous coronary intervention (PCI).

The primary aim of this pilot trial is to investigate the recruitment rate feasibility and safety of undertaking a randomised trial of simple intracoronary coronary cooling and dilution through the guiding catheter during primary PCI for STEMI to reduce myocardial infarction size.

The secondary aims are as follows:

1. The study will explore the invasive haemodynamic assessment of coronary flow and microvascular function
2. The study will explore blood biomarkers before and after treatment for myocardial infarction
3. The study will explore myocardial salvage after treatment for myocardial infarction with magnetic resonance imaging (MRI) and subsequent final infarct size.

Patients will be randomised 1:1 in the catheterisation lab when coronary angiography has demonstrated a target lesion with proposed primary PCI. Patients randomised to the intervention will receive transcatheter cooling and dilution in addition to usual clinical care. Patients randomised to control will receive usual care alone.

A combined thermistor and pressure wire Coroventis™ (Abbott Vascular) with comparable tip stiffness to standard guidewires and in routine clinical use, will be used to perform the primary PCI procedure and to measure intracoronary temperature and pressure continually throughout all procedures in all patients. This will therefore limit the procedure to a simple single wire throughout strategy in most cases. In the event that the wire fails to function properly during or after the PCI procedure it may be changed for a new wire using standard interventional techniques as appropriate

Patients randomised to intracoronary cooling and dilution(n=30), will receive an intracoronary infusion of room temperature 0.9% Normal Saline solution through the guiding catheter which will commence immediately prior to crossing the coronary occlusion with the guidewire. Using a 3-way tap in the procedural manifold an infusion pressure of 150mmHg above systolic blood pressure achieved with a pressure bag will be used to achieve a target intracoronary temperature of 6-8 C° below the baseline temperature. The infusion will continue until 10 minutes after the lesion is crossed and distal flow is restored, with only brief interruptions as required for the clinical procedure. A maximum volume of 750ml will be infused. The primary angioplasty procedure itself will be undertaken according to standard local practice. Patients randomised to the control group (n=30) will undergo primary PCI according to standard local practice.

A complete physiological study including Fractional flow reserve (FFR), resting full-cycle ratio (RFR), coronary flow reserve (CFR), resistive reserve ratio (RRR) and index of microvascular resistance (IMR) to assess microcirculation will be measured 10 minutes after reperfusion in all patients.

Patients will go on to have blood taken on the next day for the analysis of a panel of biomarkers and comparison with pre-procedure levels and in addition to have a cardiac MRI scan prior to discharge and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical ST-elevation myocardial infarction or equivalent (e.g. new onset LBBB)
* <12 Hrs after symptom onset
* Thrombolysis in myocardial infarction (TIMI) 0-1 coronary flow in a target vessel

Exclusion Criteria:

* History of severe asthma
* Pregnancy
* Severe concomitant disease or conditions with a life expectancy of less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  Patients recruited per month
Feasibility (Number of studies where all the planned measurements have been collected / total studies) | 1 year
  Number of studies where all the planned measurements have been collected / total studies
Safety (Adverse events should not be significantly higher in the treatment arm compared to control, nor plausibly caused by the treatment) | 1 year
  Adverse events should not be significantly higher in the treatment arm compared to control, nor plausibly caused by the treatment as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Index of microvascular resistance (IMR) 10 mins after completion of percutaneous coronary intervention and study infusion | 1 hour
  Distal coronary pressure during hyperaemia x mean transit time (mmHg·s)
Fractional flow reserve (FFR) 10 mins after completion of percutaneous coronary intervention and study infusion | 1 hour
  Distal coronary pressure/aortic pressure during hyperaemia
Coronary flow reserve (CFR) 10 mins after completion of percutaneous coronary intervention and study infusion | 1 hour
  Thermodilution-based ratio of hyperaemic coronary flow/basal flow
Resistive reserve ratio (RRR) 10 mins after completion of percutaneous coronary intervention and study infusion | 1 hour
  Index of microvascular resistance rest/hyperaemia
Resting full-cycle ratio (RFR) 10 mins after completion of percutaneous coronary intervention and study infusion | 1 hour
  lowest value of distal coronary pressure/aortic pressure over the entire cardiac cycle at rest
Intracoronary temperature change | 1 hour
  Intracoronary temperature change during cooling and dilution (°C)
Infusion volume | 1 hour
  Total volume of intracoronary saline infused (ml)
Infusion rate | 1 hour
  Total volume of intracoronary saline infused/infusion time (ml/min)
Chest pain during study infusion | 1 hour
  Whether new chest pain arises, or chest pain increases during study infusion
ECG changes during study infusion | 1 hour
  Amelioration or worsening of the ECG anomalies during study infusion (ST elevation/depression, T wave inversion, QT prolongation)
Heart rhythm changes during study infusion | 1 hour
  Appearance or resolution of heart rhythm disturbances during study infusion (sinus tachycardia, supraventricular tachycardia, atrial tachycardia/fibrillation/flutter, ventricular tachycardia/flutter, ventricular fibrillation, sinus bradycardia, grade I, II, or III heart block, asystole.
Myocardial blush grade 10 mins after completion of percutaneous coronary intervention and study infusion | 1 hour
  Angiographic myocardial perfusion measurement based on visual assessment of the myocardium after contrast injection. Grading: 0, no myocardial blush or contrast density; 1, minimal myocardial blush or contrast density; 2, moderate myocardial blush or contrast density but less than that obtained during angiography of a contralateral or ipsilateral non-infarct-related coronary artery; and 3, normal myocardial blush or contrast density, comparable with that obtained during angiography of a contralateral or ipsilateral non-infarct-related coronary artery
Thrombolysis in Myocardial Infarction (TIMI) flow 10 mins after completion of percutaneous coronary intervention and study infusion | 1 hour
  Visual angiographic assessment of coronary flow. Grade 0 = no perfusion; grade 1 = penetration without perfusion; 2 = partial perfusion; 3 = complete perfusion
ST segment resolution 10 mins after completion of percutaneous coronary intervention and study infusion | 1 hour
  Null, partial, or complete resolution of the ST elevation
Heart Rhythm disturbance from baseline to 12 hours | 12 hours
  Appearance or resolution of heart rhythm disturbances in the 12 hours after the procedure (sinus tachycardia, supraventricular tachycardia, atrial tachycardia/fibrillation/flutter, ventricular tachycardia/flutter, ventricular fibrillation, sinus bradycardia, grade I, II, or III heart block, asystole.
Haemodynamic compromise from baseline to 12 hours | 12 hours
  Society for Cardiovascular Angiography and Interventions (SCAI) class B or above
Left ventricular ejection fraction (LVEF) at 48 hours | 2 days
  Simpson biplane (diastolic-systolic)/diastolic left ventricular volume on echocardiography
Left ventricular ejection fraction (LVEF) at 6 months | 6 months
  Simpson biplane (diastolic-systolic)/diastolic left ventricular volume on echocardiography
Wall motion score index (WMSI) at 48 hours | 48 hours
  The wall motion score index (WMSI) is an echocardiographic parameter that numerically sums the average scores for all left ventricular segments into a single parameter and then dividing by the number of segments. 1 Normal motion; 2 = hypokinesia; 3 = akinesia; 4 = dyskinesia.
Wall motion score index (WMSI) at 6 months | 6 months
  The wall motion score index (WMSI) is an echocardiographic parameter that numerically sums the average scores for all left ventricular segments into a single parameter and then dividing by the number of segments. 1 Normal motion; 2 = hypokinesia; 3 = akinesia; 4 = dyskinesia.
Global longitudinal strain (GLS) at 48 hours | 48 hours
  Echocardiographic speckle-tracking imaging that measures the systolic shortening of left ventricular segments as percentage of their diastolic length
Global longitudinal strain (GLS) at 6 months | 6 months
  Echocardiographic speckle-tracking imaging that measures the systolic shortening of left ventricular segments as percentage of their diastolic length
Length of stay | 3-5 days
  Duration of hospital length of stay
Peak high-sensitivity cardiac troponin T (hs-cTnT, ng/l) | 1-3 days
  Myocardial injury marker. Highest hs-cTnT measurement during hospital stay
N-terminal pro-brain natriuretic peptide (NT-proBNP, ng/l) | 1-3 days
  Heart failure marker. Highest NT-proBNP measurement during hospital stay
Interleukin-1b | 1 day
  Biomarker of inflammation during myocardial infarction
Interleukin-1 receptor antagonist | 1 day
  Biomarker of inflammation during myocardial infarction
Interleukin-6 | 1 day
  Biomarker of inflammation during myocardial infarction
Interleukin-10 | 1 day
  Biomarker of inflammation during myocardial infarction
First pass microvascular obstruction extent (FP MVO) | 1-3 days
  Measured in 3 SAX levels to provide an index of %LV FP MVO
First pass microvascular obstruction extent (FP MVO) at 6 months | 6 months
  Measured in 3 SAX levels to provide an index of %LV FP MVO
Early MVO extent (% of LV) on 1 min post-gadolinium contrast enhanced MRI, adjusted for area at-risk | 1-3 days
  Cardiac magnetic resonance-based assessment
Early MVO extent (% of LV) on 1 min post-gadolinium contrast enhanced MRI, adjusted for area at-risk, at 6 months | 6 months
  Cardiac magnetic resonance-based assessment
Late MVO (presence / absence) on LGE | 1-3 days
  Cardiac magnetic resonance-based assessment
Late MVO (presence / absence) on LGE at 6 months | 6 months
  Cardiac magnetic resonance-based assessment
Initial infarct size (LGE) | 1-3 days
  Mass of infarcted myocardium calculated with the full-width at half-maximum method
Infarct size (LGE) at 6 months | 6 months
  Mass of infarcted myocardium calculated with the full-width at half-maximum method
Initial MSI (area-at-risk minus initial infarct size/area-at-risk) | 1-3 days
  Percentage of the area at risk (calculated with the Otsu method) that was not infarcted on late gadolinium enhancement (LGE) images using infarct size from the pre-discharge (Acute MSI)
MSI (area-at-risk minus initial infarct size/area-at-risk) at 6 months | 6 months
  Percentage of the area at risk (calculated with the Otsu method) that was not infarcted on late gadolinium enhancement (LGE) images using infarct size from the follow-up (Final MSI) magnetic resonance imaging
Left ventricular end-diastolic volume index (LVEDVI) | 1-3 days
  Cardiac magnetic resonance-based assessment
Left ventricular end-diastolic volume index (LVEDVI) at 6 months | 6 months
  Cardiac magnetic resonance-based assessment
Left ventricular end-systolic volume index (LVESVI) | 1-3 days
  Cardiac magnetic resonance-based assessment
Left ventricular end-systolic volume index (LVESVI) at 6 months | 6 months
  Cardiac magnetic resonance-based assessment
Cardiac Magnetic Resonance-based Left ventricular ejection fraction (LVEF) | 1-3 days
  Cardiac magnetic resonance-based assessment
Cardiac Magnetic Resonance-based Left ventricular ejection fraction (LVEF) at 6 months | 6 months
  Cardiac magnetic resonance-based assessment
Myocardial haemorrhage (presence/absence) | 1-3 days
  Cardiac magnetic resonance-based assessment
Myocardial haemorrhage (presence/absence) at 6 months | 6 months
  Cardiac magnetic resonance-based assessment
Myocardial haemorrhage extent (% of LV) | 1-3 days
  Cardiac magnetic resonance-based assessment
Myocardial haemorrhage extent (% of LV) at 6 months | 6 months
  Cardiac magnetic resonance-based assessment
Composite of all-cause mortality and hospitalization for heart failure at 6 weeks | 6 weeks
  Composite of all-cause mortality and hospitalization for heart failure at 6 weeks
Hospitalization for heart failure at 6 weeks | 6 weeks
  Hospitalization for heart failure at 6 weeks
Cardiovascular mortality at 6 weeks | 6 weeks
  Cardiovascular mortality at 6 weeks
All-cause mortality at 6 weeks | 6 weeks
  All-cause mortality at 6 weeks
Hospitalization for heart failure at 6 months | 6 months
  Hospitalization for heart failure at 6 months
Cardiovascular mortality at 6 months | 6 months
  Cardiovascular mortality at 6 months
Composite of all-cause mortality and hospitalization for heart failure at 6 months | 6 months
  Composite of all-cause mortality and hospitalization for heart failure at 6 months
All-cause mortality at 6 months | 6 months
  All-cause mortality at 6 months
Composite of all-cause mortality and hospitalization for heart failure at 12 months | 12 months
  Composite of all-cause mortality and hospitalization for heart failure at 12 months
Hospitalization for heart failure at 12 months | 12 months
  Hospitalization for heart failure at 12 months
Cardiovascular mortality at 12 months | 12 months
  Cardiovascular mortality at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Miles C Dalby, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Harefield Hospital, Uxbridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Otterspoor LC, Van 't Veer M, Van Nunen LX, Brueren GRG, Tonino PAL, Wijnbergen IF, Helmes H, Zimmermann FM, Van Hagen E, Johnson NP, Pijls NHJ. Safety and feasibility of selective intracoronary hypothermia in acute myocardial infarction. EuroIntervention. 2017 Dec 8;13(12):e1475-e1482. doi: 10.4244/EIJ-D-17-00240. PMID 28829744
- [Background] McGarvey M, Ali O, Iqbal MB, Ilsley C, Wong J, Di Mario C, Redwood S, Patterson T, Pennell DJ, Rogers P, Dalby M; ORCA-3 For the Optimal Restoration of Cardiac Activity (ORCA) Group. A feasibility and safety study of intracoronary hemodilution during primary coronary angioplasty in order to reduce reperfusion injury in myocardial infarction. Catheter Cardiovasc Interv. 2018 Feb 1;91(2):234-241. doi: 10.1002/ccd.27136. Epub 2017 Jun 21. PMID 28636165
- [Background] Erlinge D, Gotberg M, Lang I, Holzer M, Noc M, Clemmensen P, Jensen U, Metzler B, James S, Botker HE, Omerovic E, Engblom H, Carlsson M, Arheden H, Ostlund O, Wallentin L, Harnek J, Olivecrona GK. Rapid endovascular catheter core cooling combined with cold saline as an adjunct to percutaneous coronary intervention for the treatment of acute myocardial infarction. The CHILL-MI trial: a randomized controlled study of the use of central venous catheter core cooling combined with cold saline as an adjunct to percutaneous coronary intervention for the treatment of acute myocardial infarction. J Am Coll Cardiol. 2014 May 13;63(18):1857-65. doi: 10.1016/j.jacc.2013.12.027. Epub 2014 Feb 5. PMID 24509284